CLINICAL TRIAL: NCT03783104
Title: A Randomised Controlled Trial to Compare Two Different Doses of Maternal B12 Supplementation in Improving Infant B12 Deficiency and Neurodevelopment
Brief Title: Maternal B12 Supplementation to Improve Infant B12 Deficiency and Neurodevelopment
Acronym: MATCOBIND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Sitaram Bhartia Institute of Science and Research (Other); Paropakar Maternity and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13795/001
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Child Developmental Delay; Child Malnutrition; Maternal Exposure; Vitamin B 12 Deficiency
Keywords: Vitamin B12; Maternal nutrition; Neurodevelopment; Supplementation
MeSH Terms: conditions — Learning Disabilities; Child Nutrition Disorders; Vitamin B 12 Deficiency

STUDY DESIGN:
Intervention Model Description: A total of 720 recruited mothers across India and Nepal will be randomly allocated to 2 equal groups (360 each). Group 1 (Intervention) will receive 250μg of vitamin B12 supplementation delivered daily to the mother from 12 weeks gestation up to 6 months post-partum. Group 2 (Control) will receive 50μg of vitamin B12 supplementation delivered daily to the mother from 12 weeks gestation up to 6 months post-partum.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 250μg of vitamin B12 supplementation (Experimental): Group 1 (Intervention) will receive 250μg of vitamin B12 supplementation delivered daily to the mother from 12 weeks gestation up to 6 months post-partum.
  Interventions: Dietary Supplement: B12 Supplement
- 50μg of vitamin B12 supplementation (Active Comparator): Group 2 (Control) will receive 50μg of vitamin B12 supplementation delivered daily to the mother from 12 weeks gestation up to 6 months post-partum.
  Interventions: Dietary Supplement: B12 Supplement

INTERVENTIONS:
Dietary Supplement: B12 Supplement — Differential doses of vitamin B 12 supplementation in a two-armed randomised controlled trial

SUMMARY:
Vitamin B12 plays a key role in the development and normal functioning of the brain and nervous system. Unborn and new-born infants derive their vitamin B12 stores almost entirely from maternal B12 stores. As such, infants who are born to vegetarian mothers and exclusively breast fed are at a high-risk of B12 deficiency. This is because the best sources of vitamin B12 are found in animal based or fortified foods (e.g. cheese, milk and eggs). Vitamin B12 deficiency is widely reported among antenatal mothers and children, particularly in Low and Middle Income Countries (LMICs) where these food sources are uncommon.

So far, studies have shown that antenatal vitamin B12 deficiency in mothers may be associated with poorer neurodevelopment in their children. Furthermore, vitamin B12 supplementation during pregnancy and early lactation has been shown to increase maternal, breast milk, and infant levels of vitamin B12. Although existing literature documents several studies on maternal vitamin B12 supplementation, there is a lack of research on the causative effect of maternal vitamin B12 supplementation on infant development. This project, funded by the Medical Research Council (MRC), will undertake a multi-centric nutritional trial in Nepal and India, as these are two LMICs where high incidence of vitamin B12 deficiency is reported.

DETAILED DESCRIPTION:
The project is a multi-centric, double-blind and parallel two-armed randomised controlled trial divided into two stages:

Stage 1:

A total of 720 recruited mothers across India and Nepal will be randomly allocated to 2 equal groups (360 each). The patients, recruiters, developmental therapists, the laboratory and the data analyst will be blinded to the randomization code for the duration of the trial. To ensure blinding and allocation concealment, maternal supplements will be numbered sequentially outside the trial sites by a neutral party using the randomization code supplied by an offsite statistician. Group 1 (Intervention) will receive 250μg of vitamin B12 supplementation delivered daily to the mother from 12-weeks' gestation up to 6-months post-partum. Group 2 (Control) will receive 50μg of vitamin B12 supplementation delivered daily to the mother from 12-weeks' gestation up to 6- months post-partum. The mother's profile will be recorded, including information on: age, height, weight, ethnicity, education, socioeconomic status, maternal dietary assessment and intake of any supplements. Mother's blood levels for vitamin B12 status and other deficiencies will also be recorded.

Within 48 hours enrolment women will be contacted as a part of follow-up. Relevant elements of the clinical records including maternal weight, blood pressure, foetal growth and position and reports of any screening tests for congenital infections/ chromosomal anomalies will be recorded. Any acquired morbidity (including gestational diabetes, pregnancy induced hypertension, and hypothyroidism) during the period from the last visit will be noted. Any drugs or medicines started by the mother will be recorded. Both study sites will promote exclusive breastfeeding by preparing the mothers for breastfeeding in the antenatal period using structured counselling sessions led by an obstetrician or a specified health educator.

Stage 2:

The birth and post-delivery course of the new-born during hospital stay will be assessed by the medical officer and/or paediatrician for any morbidity potentially influencing neurodevelopment, such as growth retardation, congenital anomalies, seizures, neurological problems, hypoglycemia, hypothermia, hearing deficits, vision and heart disease.

After discharge, all neonates will be routinely followed with preventive and vaccination care as per standard protocols. As part of routine care, all new-borns will be screened for metabolic disorders at 7-14 days.

During routine visits, anthropometric measurements including weight, length and head circumference will be recorded and signs of micronutrient deficiency (especially anaemia and rickets) will be noted. The child care teams at both sites will encourage the initiation and establishment of exclusive breastfeeding while minimizing the use of formula feeds by providing support and counselling during hospital stay. Maternal and infant tolerance for the supplementation including any gastrointestinal symptoms will be recorded at each visit. Supplementation of the mother in both groups will be stopped at 6 months after childbirth. At 9 months, the neurodevelopmental, complementary feeding practices and home environment will be assessed and infant vitamin B12 status will be determined.

Data will be checked and encrypted after removing any "patient identifiable information". These data will be sent with the group coding sheet to a statistician blinded to intervention or control grouping. Data will be analysed using the neurodevelopmental scores at 9 months as the primary efficacy outcome variable. Biochemical prevalence of B12 deficiency in mothers during the first and third trimesters and infants after 9 months of birth will be analysed as the secondary outcome variables. Although no safety issues are expected, infant linear growth and incidence of adverse events will be the mainly safety outcomes. Data on maternal tolerance of B12 supplementation will also be collected. All primary analyses will be conducted on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give full consent (record if verbal consent is being used)
* First presentation of the mother to the antenatal clinic <12 weeks of gestation (mothers presenting later not included as the investigators may miss a proportion of the brain growth period)
* Vegetarian mothers (higher risk of deficiency; defined as self-reported dietary pattern that includes vegans and/or people who do eat egg and/or people who do consume milk and/or meat/fish < once a month)
* Mother is expecting singleton birth
* Living within an a-priori defined geographical area (to enhance efficiency of follow-up): Delhi - National Capital Region; Nepal - 10km radius of Paropakar Maternity & Women's Hospital, Kathmandu valley including the three districts of Kathmandu, Bhaktapur and Lalitpur.
* Is familiar with English, Hindi, or Nepalese

Exclusion Criteria:

* Younger mothers (<18 years; higher risk of neonatal morbidity)
* Maternal Age>35 years ( higher risk of neonatal morbidity)
* Mothers already on medicinal B12 supplementation including as B-complex or multivitamins (confounder)
* Women with multiple gestation, those diagnosed with chronic medical conditions (diabetes mellitus, hypertension, heart disease, neurological disease or thyroid disease), and those who tested positive for hepatitis B, HIV or syphilis (associated with prematurity, intrauterine growth restriction (IUGR) and other neonatal morbidities which could influence neurodevelopment)
* Women who anticipate moving out of the city before/ after delivery (follow-up difficult/not possible, 16% delivered outside Sitaram Bhartia Institute of Science & Research (SBISR) in earlier work done by Principle Investigator) (3)
* Women treated for infertility (higher risk of prematurity and neonatal complications
* Women with known pre-diagnosed mental health disorder including depression, drug or alcohol abuse likely to affect participation in the study
* Participation in another study within 4 weeks prior to trial start
* Allergy to B12 or another supplement constituent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women are eligible.
Enrollment: 720 (Estimated)
Dates: Start 2019-04-27 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Infant neurodevelopment | 9 months in all infant subjects
  The effect of higher dose oral maternal vitamin B12 supplementation on infant neurodevelopment as measured by Developmental Assessment Scales for Indian Infants (DASII) at age 9 months, as compared to low dose

SECONDARY OUTCOMES:
Maternal B12 status | First trimester (<12 weeks gestation) and third trimester (≥ 27 weeks)
  The change in biochemical parameters of maternal B12 status between first (<12 weeks gestation) and third trimester (≥ 27 weeks gestation) as measured by vitamin B12, homocysteine and holotranscobalamin levels
Infant B12 status | 9 months (± 2 weeks) of age after birth
  The change in biochemical parameters of infant B12 status at 9 months (± 2 weeks) after birth as compared to low dose
Hemoglobin levels and infant anthropometry | Between first and third trimester
  The change in hemoglobin levels in the mother
Hemoglobin levels and infant anthropometry | At 9 months after birth
  The change in hemoglobin levels in the infant
Hemoglobin levels and infant anthropometry | At 1, 2, 3, 4, 6 and 9 months after birth
  The change in infant anthropometry including weight, length, and head circumference (c)

OTHER OUTCOMES:
Socio-economic mediators of the relationship between maternal B12 status, supplementation and infant neurodevelopment | At study enrolment
  Income, education, profession
Effect of maternal diet | During the third trimester (27 weeks of gestation)
  The effect of the intervention on maternal vitamin B12 status, infant B12 status and infant neurodevelopment
Effect of type of milk feeding on infant vitamin B12 status | At 9 months (± 2 weeks) infant age
  Assessed by measuring blood levels of B12
Effect of type of milk feeding on infant neurodevelopment | At 9 months (± 2 weeks) infant age
  Assessed using the Developmental Assessment Scales for Indian Infants (DASII)
Effect of infant complementary feeding on infant vitamin B12 status | At 9 months (± 2 weeks) infant age
  Assessed by measuring blood levels of B12
Effect of infant complementary feeding on infant neurodevelopment | At 9 months (± 2 weeks) infant age
  Assessed using the Developmental Assessment Scales for Indian Infants (DASII)
Effect of maternal iron | In first and third trimester and at 9 months (± 2 weeks) infant age
  Determining any effect of maternal iron levels in first and third trimester on the relationship between infant vitamin B12 status and infant neurodevelopment
Effect of maternal vitamin D status | In first and third trimester and at 9 months (± 2 weeks) infant age
  Determine any effect of maternal vitamin D status in first and third trimester on the relationship between infant vitamin B12 status and infant neurodevelopment

CONTACTS AND LOCATIONS:
Overall Officials: Monica Lakhanpaul, Principal Investigator — University College, London
Locations (2):
- Sitaram Bhartia Institute for Science and Research, New Delhi, India
- Paropakar Maternity and Women's Hospital, Kathmandu, Nepal